CLINICAL TRIAL: NCT04248322
Title: Qualitative Assessment of the Impact of Transcutaneous Tibial Nerve Stimulation (TTNS) on Quality of Life and Participation
Brief Title: Qualitative Assessment of the Impact of TTNS on QOL and Participation
Status: Active, not recruiting | Type: Observational
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00004862
Record Dates: First submitted 2020-01-27; First posted 2020-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Neurogenic Bladder; Urinary Retention; Urinary Tract Infections; Spinal Cord Injuries
Keywords: Quality of Life; Participation; Barrier
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Urinary Retention; Urinary Tract Infections; Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects who used TTNS: Subjects will have Neurogenic Lower Urinary Tract Dysfunction and will have participated in a study with TTNS. n=20
  Interventions: Behavioral: Semi-structured interview

INTERVENTIONS:
Behavioral: Semi-structured interview — Using iterative, semi-structured interviews or focus groups to explore the lived experience with CC and usual customary care (UCC) of catheter users with NLUTD and their caretakers to generate user-defined themes regarding bladder function and catheter-related barriers and the daily impacts on one's life.

SUMMARY:
This study through the use of semi-structured interviews or focus groups will explore the lived experience with Transcutaneous Tibial Nerve Stimulation (TTNS) with Neurogenic Lower Urinary Tract Dysfunction to generate user-defined themes regarding bladder function and catheter-related barriers and the daily impacts on one's life.

DETAILED DESCRIPTION:
Identify NLUTD user-defined themes regarding bladder function and and the daily impacts on one's life Specific Aim: Using iterative, semi-structured interviews or focus groups to explore the lived experience using TTNS neuromodulation to generate user-defined themes regarding bladder function and the daily impacts on one's life.

ELIGIBILITY:
Inclusion:

Participated in TTNS Study for 1 year.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will purposively recruit consumers Y1-Y4 to explore their experience with bladder function, as well as NLUTD-related barriers and impact on one's life. Recruitment will be guided by a random sampling of patient characteristics to promote comprehensive sampling as follows: usual bladder management, and etiology of NLUTD (n=20).
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Consumer user-defined themes from qualitative interviews | Collected once at study completion at 1 year
  Explore the lived experience using the transcutaneous tibial nerve stimulation to generate user-defined themes regarding bladder function and the daily impacts on one's life. Qualitative analysis will be used to define these themes about how TTNS impacted ones life, and bladder function

SECONDARY OUTCOMES:
Follow-up calls regarding user-defined themes | through study completion, an average of 1 year
  Possible follow-up calls for clarification on user-defined themes (primary outcome) may need to be done to

CONTACTS AND LOCATIONS:
Overall Officials: Emily Leonard, PhD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- MedStar National Rehabilitation Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No